CLINICAL TRIAL: NCT02713438
Title: Physical Activity, and Health-Related Quality of Life: Dyadic Research in the Context of Forming Individual, Dyadic, and Collaborative Plans (Trial 1: Parent-Child Dyads)
Brief Title: Effects of Individual, Dyadic, and Collaborative Plans on Physical Activity in Parent-Child Dyads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014/15/B/HS6/00923_PCD; 2014/15/B/HS6/00923 (Other Grant/Funding Number: National Science Centre, Poland)
Record Dates: First submitted 2016-03-10; First posted 2016-03-18 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Health Behavior
Keywords: Physical activity; Planning; Implementation intention; Quality of life; Body weight
MeSH Terms: conditions — Health Behavior; Motor Activity; Body Weight | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Individual Planning (Experimental): Participants are filling in the planning forms, referring to their individual physical activity. Both members of the dyad form their own, interdependent plans.
  The following behavior change techniques (BCT) are included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/coping planning. Applications of all BCT included references to planning.
  Interventions: Behavioral: Individual Planning; Behavioral: Education
- Dyadic Planning (Experimental): Participants are filling in the planning forms jointly. Planning refers to physical activity of only one person in the dyad, the child. The parent is actively participating in forming plans by the child.
  The following BCT are included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/coping planning. Applications of all BCT included references to planning.
  Interventions: Behavioral: Dyadic Planning; Behavioral: Education
- Collaborative Planning (Experimental): Participants are filling in the planning forms jointly. Planning refers to physical activity of both persons in the dyad (child and parent). Physical activity may be performed jointly by both persons in the dyad.
  The following BCT are included in the planning intervention protocol: action planning, barrier identification, prompting self-talk, relapse prevention/coping planning. Applications of all BCT included references to planning.
  Interventions: Behavioral: Collaborative Planning; Behavioral: Education
- Education (Active Comparator): The education group received extended physical activity and healthy nutrition education program. The education includes: (1) the guidelines for physical activity and healthy nutrition, tailored to age and health status of the participant, (2) the examples of exercises and their metabolic equivalent; (3) information about healthy body mass and body composition.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Individual Planning — CONTENT: The planning materials and forms have sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans. Action plans (referring to when, when, and how the individual will act) as well as coping plans (referring to how to overcome potential difficulties, risky situations or temptations to not engage in physical activity).
  Each participant forms their plans individually, without consulting the dyadic partner, but discussing the plans with the experimenter.
  Arms: Individual Planning
Behavioral: Dyadic Planning — CONTENT: The planning materials and forms have sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans. Action plans (referring to when, when, and how the individual will act) as well as coping plans (referring to how to overcome potential difficulties, risky situations or temptations to not engage in physical activity).
  Both partners in the dyad jointly form one plan. This jointly developed plan is discussed with the experimenter. The plan focuses on physical activity of only one person in the dyad: the child (parent-child dyads).
  Arms: Dyadic Planning
Behavioral: Collaborative Planning — CONTENT: The planning materials and forms have sections: (a) information on the importance of planning, including examples of how planning works and what it affects, (b) instructions of what should be included in a good plan (the when, where, and how components), (c) formulating action and coping plans. Action plans (referring to when, when, and how the individual will act) as well as coping plans (referring to how to overcome potential difficulties, risky situations or temptations to not engage in physical activity).
  Both partners in the dyad jointly form one plan. This jointly developed plan is discussed with the experimenter. The plan focuses on physical activity of both persons within the dyad (parent and child) and include some plans for joint physical activity.
  Arms: Collaborative Planning
Behavioral: Education — CONTENT: The education materials address physical activity and healthy nutrition guidelines for age groups. Participants receive a set of educational materials about types of physical activity (PA), PA intensity, exercise calorie expenditure, strength and endurance training, stretching, and general nutrition guidelines in terms of meal composition, and nutrients, meal frequency. The materials exclude any planning statements.
  The education is delivered by the experimenter to a parent-child dyad and discusses individual guidelines for both dyadic partners.

SUMMARY:
AIMS: The project aims at investigating of the effects of three types of planning (individual planning, collaborative planning, and dyadic planning) on physical activity.The influence of three planning interventions are compared with an active control condition, including physical activity education.

PARTICIPANTS: The effects of the interventions are evaluated among parent-child (aged 10-14) dyads, with a minimum of 50 dyads enrolled into the each arm of the trial (a total of 200 dyads). The interventions consist of six planning sessions.

DESIGN: The dyads are randomly assigned to one of four experimental conditions. The assessment of the main and secondary outcomes is conducted at the baseline, at 1 week after the first intervention session, at post-intervention (after six intervention sessions are completed), and at 6-, and 12-month follow-ups.

OUTCOMES: Physical activity constitutes the main outcome, whereas health-related quality of life (HRQOL), body mass index, as well as the self-regulatory strategy called the use of planning (individual, dyadic and collaborative) are secondary outcomes.

DETAILED DESCRIPTION:
Individual planning (also known as implementation intentions or action and coping planning) is a regulatory strategy, which refers to making plans on when, where, and how to perform an intended behavior. In dyadic planning, a target person is setting plans together with a partner on when, where, and how the target person will individually engage in behavior change. The concept of dyadic planning differs from the conceptualization of collaborative plans, where two individuals make plans on how to enact a behavior together.

The study will evaluate the effects of a short-term planning intervention. The intervention includes a total of six sessions: two face-to-face sessions with the experimenter (delivered over two weeks) and three sessions delivered over phone (over the following three weeks), one face-two-face session (delivered at one month after the third session delivered over the phone). The delivery has an individual format (the experimenter + the dyad). The total time from first to sixth session is 2 months. The setting for the interventions will include schools (school nurse office) or/and participant's home. The same format, schedule, delivery, and setting will be used for conducting active control group procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children (age 10-14) and one healthy parents (any gender) or legal guardians
* Child or parent/legal guardian with chronic conditions but without contraindications for moderate intensity physical activity

Exclusion Criteria:

* Children younger than 10 years old
* Parents who declared plans for changing residence during the following year (e.g., due to moving to another region of the country)
* No parental consent at the baseline
* No child consent at the baseline
* Existing diseases with contraindications for moderate intensity physical activity

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2023-11 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Physical activity | Change from the baseline physical activity at 8 months
  Accelerometry: ActiGraph (the model: wGT3X-B)

SECONDARY OUTCOMES:
Health-related quality of life (HRQOOL) | Change from baseline HRQOL at 8 months
  WHOQOL-BREF (Skevington et al., 2004), the measure HRQOL among adults (parents)
Health-related quality of life (HRQOL) | Change from baseline HRQOL at 8 months
  KIDSCREEN-10 (Ravens-Sieberer et al., 2010); the measure HRQOL among children
The use of planning | Change from baseline use of planning at 2 months
  The self-reported use of planning (individual, dyadic and collaborative) questionnaire, based on Luszczynska (2006)
Body mass index (BMI) | Change from baseline BMI at 8 months
  Certified and standardized body weight scales (Beurer; European Union safety certificate; measurement error < 5%) and measuring rods will be used. BMI will be calculated as body weight (in kilograms) divided by a square height (in meters)
Physical activity behavior | Baseline (before the intervention) to 1 week after the first face-to face intervention session); Baseline to 6-month follow-up
  The International Physical Activity Questionnaire (IPAQ) (Craig et al., 2003); open-ended questions indicating the minutes and the number of occasions of physical activity behavior per week; higher scores represent better outcome
Sedentary behavior | Baseline (before the intervention) to 1 week after the first face-to face intervention session); Baseline to 6-month follow-up
  Accelerometry: ActiGraph (the model: wGT3X-B)

OTHER OUTCOMES:
Habitual physical activity | Change from baseline habitual physical activity at 8 months
  Self-reported habit index (physical activity) questionnaire (Gardner et al., 2012)
Habitual sedentary behavior | Change from baseline habitual sedentary behavior at 8 months
  Self-reported habit index (sedentary behavior) questionnaire (Gardner et al., 2012)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Luszczynska, PhD, Principal Investigator — SWPS University of Social Sciences and Humanities
Locations (1):
- University of Social Sciences and Humanities, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data will be made publicly available in 3 years after the completion of the trial

REFERENCES:
- [Background] Burkert S, Knoll N, Luszczynska A, Gralla O. The interplay of dyadic and individual planning of pelvic-floor exercise in prostate-cancer patients following radical prostatectomy. J Behav Med. 2012 Jun;35(3):305-17. doi: 10.1007/s10865-012-9416-2. Epub 2012 Mar 28. PMID 22454228
- [Background] Prestwich A, Conner MT, Lawton RJ, Ward JK, Ayres K, McEachan RR. Randomized controlled trial of collaborative implementation intentions targeting working adults' physical activity. Health Psychol. 2012 Jul;31(4):486-95. doi: 10.1037/a0027672. Epub 2012 Apr 2. PMID 22468716
- [Background] Luszczynska A. An implementation intentions intervention, the use of a planning strategy, and physical activity after myocardial infarction. Soc Sci Med. 2006 Feb;62(4):900-8. doi: 10.1016/j.socscimed.2005.06.043. Epub 2005 Aug 10. PMID 16095786
- [Background] Ravens-Sieberer U, Erhart M, Rajmil L, Herdman M, Auquier P, Bruil J, Power M, Duer W, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; European KIDSCREEN Group. Reliability, construct and criterion validity of the KIDSCREEN-10 score: a short measure for children and adolescents' well-being and health-related quality of life. Qual Life Res. 2010 Dec;19(10):1487-500. doi: 10.1007/s11136-010-9706-5. Epub 2010 Jul 30. PMID 20668950
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Hagger MS, Luszczynska A. Implementation intention and action planning interventions in health contexts: state of the research and proposals for the way forward. Appl Psychol Health Well Being. 2014 Mar;6(1):1-47. doi: 10.1111/aphw.12017. Epub 2013 Oct 8. PMID 24591064
- [Background] Sniehotta FF, Scholz U, Schwarzer R. Action plans and coping plans for physical exercise: A longitudinal intervention study in cardiac rehabilitation. Br J Health Psychol. 2006 Feb;11(Pt 1):23-37. doi: 10.1348/135910705X43804. PMID 16480553
- [Background] Burkert S, Scholz U, Gralla O, Roigas J, Knoll N. Dyadic planning of health-behavior change after prostatectomy: a randomized-controlled planning intervention. Soc Sci Med. 2011 Sep;73(5):783-92. doi: 10.1016/j.socscimed.2011.06.016. Epub 2011 Jul 12. PMID 21807446
- Available data/document: Study Protocol — https://drive.google.com/file/d/1bosgzFmvKglMyMjhELiSg-fqzw1pn1nf/view?usp=sharing — The handbook with the protocol for experimenters (in English)